CLINICAL TRIAL: NCT00980031
Title: Aldosterone Blockade to Prevent Myocardial Remodeling In Patients With Controlled Essential Hypertension
Acronym: Aldosterone
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ended prior to study completion
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 07-14634
Record Dates: First submitted 2009-09-11; First posted 2009-09-18 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Myocardial Remodeling
Keywords: Aldosterone Blockade; Aldosterone Receptor Blockers; cardiac chamber size; wall thickness; left ventricular ejection fraction; left atrial volumes; diastolic function
MeSH Terms: interventions — Eplerenone; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactose Tablet (Placebo Comparator): Compounded capsule using Lactose Monohydrate Powder
  Interventions: Drug: Lactose Tablet
- Eplerenone (Active Comparator): 25 mg tablet placed in a capsule filled with Lactose Monohydrate Powder.
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — 25mg PO daily (QD)for 6 months
  Other Names: Inspra
  Arms: Eplerenone
Drug: Lactose Tablet — Lactose tablet
  Arms: Lactose Tablet

SUMMARY:
The goal of this project is to investigate the effects that the addition of aldosterone blockade with eplerenone will have on the progression of diastolic dysfunction in patients with controlled essential hypertension.

DETAILED DESCRIPTION:
The purpose of this project is to determine if eplerenone, an aldosterone blocker, prevents remodelling of the heart in patients with controlled essential hypertension, defined as having a blood pressure of equal to or less than 130/80 in diabetics and equal to or less than 140/90 in non-diabetics. This study will investigate if the addition of 25 milligrams of eplerenone daily to a subject's hypertension medication regimen will prevent the progression or development of diastolic dysfunction. Echocardiography will be used to measure the changes in heart structure of subjects receiving eplerenone versus subjects receiving placebo (a drug that may resemble the study drug but contains no active ingredient). Approximately 30 subjects will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

* Treated and controlled hypertension
* Less than 140/90 in non-diabetics
* Less than 130/80 in diabetics

Exclusion Criteria:

* currently receiving an aldosterone blocker
* clinical evidence of congestive heart failure
* prior myocardial infarction
* renal dysfunction with a creatinine clearance of less than 40ml/min
* serum potassium > 5.5meq/L at initiation
* concomitant use of a medication that inhibits the CYP3A4 enzyme (ketoconazole, itraconazole, nefazodone, troleandomycin, clarithromycin, ritonavir, nelfinavir)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Myocardial Remodeling (cardiac chamber sizes, wall thickness, left ventricular ejection fraction, left atrial volumes, and diastolic function) assessed by transthoracic echocardiogram | 6 months

SECONDARY OUTCOMES:
Blood Pressure | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: M Jeff Holmberg, MD, PhD, Principal Investigator — Creighton Cardiology
Locations (1):
- Creighton University Medical Center (including ambulatory centers), Omaha, Nebraska, United States